CLINICAL TRIAL: NCT01964261
Title: A Feasibility Study of the Ability of the Neural Prosthetic System 2 to Provide Direct Closed Loop Cortical Control of Extracorporeal Devices Through the Use of Intracortical Microstimulation in Patients With Quadriplegia
Brief Title: Sensory Motor Transformations in Human Cortex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richard A. Andersen, PhD (Other)
Collaborators: University of Southern California (Other); Rancho Los Amigos National Rehabilitation Center (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Richard A. Andersen, PhD, James G. Boswell Professor of Neuroscience, California Institute of Technology
Organization: California Institute of Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS-13-00492
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Quadriplegia
Keywords: Neural; Prosthetic; Brain machine interface; brain computer interface; brain control; paralysis; tetraplegia; quadriplegia; spinal cord injury; stimulation; sensory feedback
MeSH Terms: conditions — Quadriplegia; Paralysis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neural Prosthetic System 2 (Experimental): The Neural Prosthetic System 2 consists of three Neuroport Arrays, which are described in detail in the intervention description. Two of the three Neuroport Arrays are inserted into the posterior parietal cortex, an area of the brain used in reach and grasp planning. The third Neuroport Array is inserted into somatosensory cortex, specifically S1 which represents sensory feedback for the hand and fingers. The arrays are inserted and the percutaneous pedestal is attached to the skull during a surgical procedure. Following surgical recovery the subject will participate in study sessions 3-5 times per week in which they will learn to control an end effector by thought augmented with sensory feedback via intracortical microstimulation. They will then use the end effector to perform various reach and grasp tasks.
  Interventions: Device: Neural Prosthetic System 2 (NPS2)

INTERVENTIONS:
Device: Neural Prosthetic System 2 (NPS2) — The NPS2 comprises 3 NeuroPort Arrays (SIROF). The tip of the electrodes are sputtered iridium oxide film (SIROF). Each array is comprised of 100 1.5 mm microelectrodes organized on a 4mm x 4mm silicon base that is 0.25 mm thick. Each microelectrode is insulated with Parylene-C polymer and is electrically isolated from neighboring electrodes by non-conducting glass. Of the 100 electrodes, 96 are wire bonded using 25m gold alloy insulated wires sealed with a silicone elastomer. The wire bundle is potted to a printed circuit board with epoxy, the circuit board is inserted into the Patient Pedestal (percutaneous connector), and then the Patient Pedestal is filled with silicone elastomer. Two fine platinum reference wires are also attached to the Patient Pedestal. The Patient Pedestal is 19 mm wide at the skin interface.
  Other Names: NeuroPort Array

SUMMARY:
This research study is being conducted to develop a brain controlled medical device, called a brain-machine interface. The device will provide people with a spinal cord injury some ability to control an external device such as a computer cursor or robotic limb by using their thoughts along with sensory feedback.

Development of a brain-machine interface is very difficult and currently only limited technology exists in this area of neuroscience. Other studies have shown that people with high spinal cord injury still have intact brain areas capable of planning movements and grasps, but are not able to execute the movement plans. The device in this study involves implanting very fine recording electrodes into areas of the brain that are known to create arm movement plans and provide hand grasping information and sense feeling in the hand and fingers. These movement and grasp plans would then normally be sent to other regions of the brain to execute the actual movements. By tying into those pathways and sending the movement plan signals to a computer instead, the investigators can translate the movement plans into actual movements by a computer cursor or robotic limb.

A key part of this study is to electrically stimulate the brain by introducing a small amount of electrical current into the electrodes in the sensory area of the brain. This will result in the sensation of touch in the hand and/or fingers. This stimulation to the brain will occur when the robotic limb touches the object, thereby allowing the brain to "feel" what the robotic arm is touching.

The device being used in this study is called the Neuroport Array and is surgically implanted in the brain. This device and the implantation procedure are experimental which means that it has not been approved by the Food and Drug Administration (FDA). One Neuroport Array consists of a small grid of electrodes that will be implanted in brain tissue and a small cable that runs from the electrode grid to a small hourglass-shaped pedestal. This pedestal is designed to be attached to the skull and protrude through the scalp to allow for connection with the computer equipment. The top portion of the pedestal has a protective cover that will be in place when the pedestal is not in use. The top of this pedestal and its protective cover will be visible on the outside of the head. Three Neuroport Arrays and pedestals will be implanted in this study so three of these protective covers will be visible outside of the head. It will be possible to cover these exposed portions of the device with a hat or scarf.

The investigators hope to learn how safe and effective the Neuroport array plus stimulation is in controlling computer generated images and real world objects, such as a robotic arm, using imagined movements of the arms and hands.

DETAILED DESCRIPTION:
The long-term objective of this application is to understand cortical processing of sensory to motor transformations within the human cerebral cortex. A vast number of computations must be performed to achieve sensory-guided motor control. Standing out among these computations, visual information of the goals of action must be transformed from the coordinates of the retina to the coordinates of effectors used for movement, for instance limb coordinates for reaching under visual guidance and to world coordinates for interactions in the environment. Once an object is grasped, somatosensory signals from the hand are required for dexterous manipulation of grasped objects. Internal models within the sensory motor pathway are essential for estimating the current state of the body and the external environment, accounting for lags in sensory feedback, and calibrating the body to the environment.

We will use the rare opportunity of being able to record from populations of single neurons in a clinical study designed to develop neural prosthetics for tetraplegic participants paralyzed by spinal cord injuries. Cortical implants of microelectrode arrays will be made within three key locations in the sensorimotor system: primary motor cortex, primary somatosensory cortex, and posterior parietal cortex. These microelectrode arrays enable both recording and intracortical microstimulation.

We will test the hypothesis that somatosensory and motor cortex represent imagined reaches in hand coordinates, but posterior parietal cortex is task dependent, and it's population neural activity can flexibly change coordinate frames depending on the effector used in the task. Percepts evoked by intracortical microstimulation and imagined sensations will be used to understand the representation of cutaneous and proprioceptive information within primary somatosensory cortex and posterior parietal cortex. The hypothesis to be tested is that imagined sensation and electrically evoked sensations are highly overlapping - not just in primary somatosensory cortex but also in posterior parietal cortex. Lastly, we hypothesize that the posterior parietal cortex contains in humans an internal model of state estimation that shows plasticity for both natural and brain-control behaviors and transfers this learning to motor cortex.

These studies will not only greatly advance our understanding of the human sensorimotor cortical circuit, but also will provide basic knowledge for the design of future neural prosthetics.

ELIGIBILITY:
Inclusion Criteria:

* High cervical spinal lesion
* Age 22-65
* Able to provide informed consent
* Able to understand and comply with instructions in English
* Communicate via speech
* Surgical clearance
* Life expectancy greater than 12 months
* Travel up to 60 miles to study locations up to five days per week
* Caregiver monitor for surgical site complications and behavioral changes on a daily basis
* Psychosocial support system

Exclusion Criteria:

* Presence of memory problems
* Intellectual impairment
* Psychotic illness or chronic psychiatric disorder, including major depression if untreated
* Poor visual acuity
* Pregnancy
* Active infection or unexplained fever
* Scalp lesions or skin breakdown
* HIV or AIDS infection
* Active cancer or chemotherapy
* Diabetes
* Autonomic dysreflexia
* History of seizure
* Implanted hydrocephalus shunt
* Previous neurosurgical history affecting parietal lobe function
* Medical conditions contraindicating surgery and chronic implantation of a medical device
* Prior cranioplasty
* Unable to undergo MRI or anticipated need for MRI during study
* Nursing an infant or unwilling to bottle-feed infant
* Chronic oral or intravenous use of steroids or immunosuppressive therapy
* Suicidal ideation
* Drug or alcohol dependence
* Planning to become pregnant, or unwilling to use adequate birth control
* Implanted Cardiac Defibrillator, Pacemaker, vagal nerve stimulator, or spinal cord stimulator.
* Implanted deep brain stimulator (DBS), DBS leads, or cochlear implant.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2013-11-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient control over the end effector (virtual or physical) | Nine years after array implantation
  The primary effectiveness objective of this study is to evaluate the effectiveness of the NPS2 in controlling virtual or physical end effectors. Signals from posterior parietal cortex will allow the subject to control the end effector with accuracy significantly greater than chance; the subject will be able to perceive and discriminate ICMS above the level of chance; and,incorporating stimulation will improve the subject's control over the end effector.
  We will evaluate the effectiveness of the NPS2 primarily by calculating the accuracy of the subjects' control over the end effector with and without ICMS, and comparing these different accuracies to the chance level, and to each other. Each subject will serve as his or her own control.
Absence of infection or irritation | Nine years after array implantation
  The primary objective of this study is to evaluate the safety of the NPS2. Implantation will not be associated with infection or irritation, and that the serious adverse event rate will not rise above 1%. We will evaluate the safety of the NPS2 by inspecting the subjects' scalps for evidence of reddening or discharge, by performing regularly scheduled neurologic history and physical exam, and by obtaining feedback from the subjects. The condition of the area will be compared with its condition on previous visits, history will be obtained regarding new symptoms and neurological and physical exam will be compared to baseline exams.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Andersen, PhD, Principal Investigator — California Institute of Technology; Charles Liu, MD, PhD, Principal Investigator — University of Southern California, Rancho Los Amigos Rehabilitation Center; Dan Kramer, MD, Principal Investigator — University of Colorado, Denver; Luke Bashford, PhD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Southern California, Los Angeles, California
  - Richard Andersen, Pasadena, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado

REFERENCES:
- [Derived] Bashford L, Rosenthal IA, Kellis S, Bjanes D, Pejsa K, Brunton BW, Andersen RA. Neural subspaces of imagined movements in parietal cortex remain stable over several years in humans. J Neural Eng. 2024 Aug 28;21(4):046059. doi: 10.1088/1741-2552/ad6e19. PMID 39134021
- [Derived] Armenta Salas M, Bashford L, Kellis S, Jafari M, Jo H, Kramer D, Shanfield K, Pejsa K, Lee B, Liu CY, Andersen RA. Proprioceptive and cutaneous sensations in humans elicited by intracortical microstimulation. Elife. 2018 Apr 10;7:e32904. doi: 10.7554/eLife.32904. PMID 29633714